CLINICAL TRIAL: NCT00557570
Title: Clinical, Virologic, and Immunologic Evaluation and Monitoring of Patients With Known or Suspected HIV Infection
Brief Title: Evaluation and Monitoring of Patients With HIV Infectionn
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 950072; 95-I-0072
Record Dates: First submitted 2007-11-10; First posted 2007-11-14 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2009-10-29

CONDITIONS: HIV
Keywords: Antiretroviral; Opportunistic Infection; treatment experienced; treatment naive
MeSH Terms: conditions — Opportunistic Infections

SUMMARY:
This study is designed to learn more about HIV infection and the conditions associated with it.

Patients 18 years of age or older with known or suspected HIV infection may be eligible for this study. Patients may have participated in previous NIH studies.

Participants will have periodic physical examinations and blood tests, including evaluations for responses to treatment. Treatment consistent with accepted standard medical practice will be individualized for each patient. Patients who previously participated in a NIH study will be followed for possible long-term benefits or side effects of treatment. Patients treated with alpha-interferon or interleukin-2 (IL-2) may continue treatment with that medication if it is felt that they might benefit from it. Blood samples may be drawn as part of standard medical care and for research purposes. Other tests may be done as appropriate for diagnosis and treatment, including, for example, a chest X-ray, electrocardiogram, or tissue biopsy. Patients will be seen for follow-up visits at regular intervals to monitor treatment progress.

Certain patients currently enrolled in a NIH study of IL-2 treatment may participate in a phase of the study that adds a corticosteroid, such as hydrocortisone, prednisone, or prednisonolone, to the regimen. Patients whose CD4 counts did not increase with IL-2 will receive corticosteroids (by mouth or by vein) in an open manner. Patients who responded to IL-2 therapy will be randomly assigned to receive corticosteroids or a placebo (inactive substance) during IL-2 infusions in a blinded manner, so that neither the patient nor the medical staff will know which patients are receiving the drug and which are receiving a placebo. Participants will be requested to receive at least three rounds of treatment with corticosteroid or placebo.

Patients currently taking IL-2 by subcutaneous injection (under the skin) may participate in an optional part of the study to receive future IL-2 cycles at home instead of at or near the Clinical Center. Patients who have shown an ability to self-administer and tolerate IL-2 injections with minimal supervision and minimal side effects may be eligible for this option. Home administration of IL-2 involves less frequent data and safety monitoring, and no on-site medical evaluation at the very beginning of each cycle. Participants will continue to be seen at the Clinical Center for regularly scheduled follow-up visits and medical evaluations before the start of each IL-2 cycle to determine if it is safe to begin that cycle. Patients will have a case manager who will place monitoring calls on days 2 and 4 of the cycle and a third follow-up call 1 week later. Patients will be responsible for contacting a study staff member if complications of other problems develop at other times.

DETAILED DESCRIPTION:
This study is designed as a prospective, observational and treatment study, with ongoing monitoring of the progression of HIV infection and HIV-related disease processes. A data base, not otherwise obtainable, will be collected of unusual disease processes related to HIV infection, and of the long-term effects of experimental treatments that patients may have received under earlier protocols for HIV and related infections. Up to 500 patients with known or suspected HIV-infection will be enrolled. Minimal studies scheduled for each visit will include monitoring of immune status, routine safety laboratory tests, and evaluation for possible opportunistic infections. Treatment plans will be individualized for each patient's particular condition, and the number and length of additional visits and diagnostic evaluations will vary accordingly. Specific treatment regimens will be in accordance with standard medical practice.

ELIGIBILITY:
* INCLUSION CRITERIA:

HIV-infection, as documented by positive HIV ELISA and Western Blot. Patients may also be included if they have laboratory or clinical evidence suggestive of possible HIV-infection.

Age 18 years or older.

Ability to give written, informed consent.

CD4 cell count of any level.

Patients may be receiving anti-retroviral therapy, and any medications provided by their primary physician for the treatment of HIV and its complications.

Patients who lack primary medical care outside the NIH may be enrolled in this protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600
Dates: Start 1995-02-11; Primary Completion 2009-10-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Kopp JB, Miller KD, Mican JA, Feuerstein IM, Vaughan E, Baker C, Pannell LK, Falloon J. Crystalluria and urinary tract abnormalities associated with indinavir. Ann Intern Med. 1997 Jul 15;127(2):119-25. doi: 10.7326/0003-4819-127-2-199707150-00004. PMID 9230000
- [Background] Gea-Banacloche JC, Weiskopf EE, Hallahan C, Lopez Bernaldo de Quiros JC, Flanigan M, Mican JM, Falloon J, Baseler M, Stevens R, Lane HC, Connors M. Progression of human immunodeficiency virus disease is associated with increasing disruptions within the CD4+ T cell receptor repertoire. J Infect Dis. 1998 Mar;177(3):579-85. doi: 10.1086/514233. PMID 9498435
- [Background] Andrieu JM, Lu W, Levy R. Sustained increases in CD4 cell counts in asymptomatic human immunodeficiency virus type 1-seropositive patients treated with prednisolone for 1 year. J Infect Dis. 1995 Mar;171(3):523-30. doi: 10.1093/infdis/171.3.523. PMID 7876597
- [Derived] Mahnke YD, Greenwald JH, DerSimonian R, Roby G, Antonelli LR, Sher A, Roederer M, Sereti I. Selective expansion of polyfunctional pathogen-specific CD4(+) T cells in HIV-1-infected patients with immune reconstitution inflammatory syndrome. Blood. 2012 Mar 29;119(13):3105-12. doi: 10.1182/blood-2011-09-380840. Epub 2012 Jan 4. PMID 22219223
- [Derived] Antonelli LR, Mahnke Y, Hodge JN, Porter BO, Barber DL, DerSimonian R, Greenwald JH, Roby G, Mican J, Sher A, Roederer M, Sereti I. Elevated frequencies of highly activated CD4+ T cells in HIV+ patients developing immune reconstitution inflammatory syndrome. Blood. 2010 Nov 11;116(19):3818-27. doi: 10.1182/blood-2010-05-285080. Epub 2010 Jul 26. PMID 20660788